CLINICAL TRIAL: NCT01125748
Title: A Phase IV, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Persistency of Response With or Without Xolair After Long-term Therapy (XPORT)
Brief Title: A Study Evaluating the Persistency of Response With or Without Xolair (Omalizumab) After Long-term Therapy
Acronym: XPORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q4777n; ML01347 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-05-14; First posted 2010-05-18 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Omalizumab (Experimental): Participants received omalizumab subcutaneously at the same dose and dosing interval as administered prior to enrollment in this study. The dose of omalizumab was either a minimum of 0.008 mg/kg/IgE (IU/mL) every 2 weeks or a minimum of 0.016 mg/kg/IgE (IU/mL) every 4 weeks for 48 weeks.
  Interventions: Drug: Omalizumab; Drug: Asthma therapies
- Placebo (Placebo Comparator): Participants received placebo subcutaneously at the same dosing interval as omalizumab was administered prior to enrollment in this study.
  Interventions: Drug: Placebo; Drug: Asthma therapies

INTERVENTIONS:
Drug: Omalizumab — Omalizumab was supplied as a sterile, white, preservative-free, lyophilized powder in single-use vials that was reconstituted with sterile water for injection.
  Other Names: Xolair
  Arms: Omalizumab
Drug: Placebo — Placebo contained the same ingredients as the omalizumab formulation, excluding omalizumab.
  Arms: Placebo
Drug: Asthma therapies — Participants could receive 1 or more of the following medications as concomitant asthma therapy: Inhaled corticosteroids; long acting beta-agonists; zafirlukast or other leukotriene receptor antagonist; zileuton or other 5-lipoxygenase enzyme inhibitors; oral, inhaled, and/or nasal anticholinergic therapy; mast-cell stabilizers; theophyllines; chronic oral corticosteroids, defined as a minimum dose of oral prednisone of 2 to 40 mg/day or 5 to 80 mg every other day.

SUMMARY:
This was a randomized, double-blind, placebo-controlled, 2-arm, 1-year study of participants who completed the EXCELS study (NCT00252135) and had received long-term treatment with Xolair. In addition, participants who did not participate in the EXCELS study but received long-term (~5 years) treatment with Xolair were allowed to enter the study.

DETAILED DESCRIPTION:
The treatment designation for participants who reached the primary efficacy endpoint (1 protocol-defined severe asthma exacerbation) was unblinded to allow appropriate clinical intervention. Participants who had their treatment designation unblinded remained in the study for ongoing evaluation of safety and were allowed to continue on study drug known to be Xolair (or to start study drug known to be Xolair if they were in the placebo group).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF). In the case of a minor, consent must be given by the child's parent or legally authorized representative.
* Participants who have completed the EXCELS study prior to this study must have met all inclusion criteria for enrollment in the EXCELS study.
* History of positive skin test or in vitro reactivity to an aeroallergen.
* Continuous Xolair (omalizumab) exposure from the beginning of the EXCELS study to randomization into this study (if the participant participated in the EXCELS study), or within the previous 5 years prior to randomization into this study (if the participant did not participate in the EXCELS study). For the purposes of this study, continuous Xolair exposure is defined as having missed no more than 25% of scheduled Xolair doses. In addition, a maximum of 2 doses can be missed within the last 6 months before being randomized into this study. For participants who did not participate in the EXCELS study, missed-dose rates will be based on their injection records.
* Patients who participated in the EXCELS study must have completed the EXCELS study and not discontinued Xolair since the completion of the EXCELS study.
* Diagnosis of moderate to severe persistent allergic asthma while on Xolair as defined per physician's assessment.
* Stable dosing of current asthma therapies, in addition to Xolair, over 2 months prior to enrollment.
* Serum IgE level ≥ 30 to ≤ 700 IU/mL before initiation of Xolair treatment (prior to the EXCELS study enrollment or earlier).
* Body weight ≥ 30 to ≤ 150 kg.
* Treatment with Xolair consistent with the US package insert (USPI) (based on the dosing table, recommended dose, administration, and dosing interval) prior to enrollment to this study.
* Participants who participated in the EXCELS study must be willing to allow their EXCELS study data to be used in this study as part of baseline demographic values (such as forced expiratory volume in 1 second [FEV1] and Asthma Control Test [ACT]), as documented in the ICF.

Exclusion Criteria:

* Participation in other therapy trials or planned participation during the following year from screening.
* Contraindication to Xolair therapy (eg, participants who experienced a severe hypersensitivity reaction to Xolair).
* Acute asthma exacerbation within the 2 months immediately prior to screening that required any of the following: Initiation of systemic corticosteroids, increased dosing of systemic corticosteroids relative to "stable" dose, doubling of inhaled corticosteroid (ICS) dosing, emergency room visit, and hospitalization.
* Any significant, or unstable, systemic disease (eg, infection, hematologic, renal, hepatic, cardiovascular diseases, or gastrointestinal diseases), or a recent hospitalization because of systemic disease within the previous 2 months.
* Diagnosis of active lung disease other than asthma.
* Having more than 10 pack-years smoking history.
* Diagnosis of cystic fibrosis.
* Use of an experimental drug within 30 days prior to study screening.
* Unable or unwilling to comply with study procedures and visits (eg, spirometry, blood draws).
* Have elevated serum IgE levels for reasons other than allergy (eg, parasite infections, hyperimmunoglobulin E syndrome, Wiskott-Aldrich syndrome, or bronchopulmonary aspergillosis).
* Pregnancy, lactation, or any planned pregnancy in the following year.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2010-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (90):
- United States (90):
  - Huntsville, Alabama
  - Little Rock, Arkansas
  - Bakersfield, California
  - Fresno, California
  - Granada Hills, California
  - Los Angeles, California
  - Napa, California
  - Redwood City, California
  - Sacramento, California
  - San Francisco, California
  - San Mateo, California
  - Studio City, California
  - Walnut Creek, California
  - Centennial, Colorado
  - Thornton, Colorado
  - Waterbury, Connecticut
  - Bay Pines, Florida
  - Clearwater, Florida
  - Loxahatchee Groves, Florida
  - Ocala, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Albany, Georgia
  - Columbus, Georgia
  - Gainesville, Georgia
  - Chicago, Illinois
  - Glen Carbon, Illinois
  - Park Ridge, Illinois
  - Fort Wayne, Indiana
  - Overland Park, Kansas
  - Topeka, Kansas
  - Lexington, Kentucky
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - Baltimore, Maryland
  - Ellicott City, Maryland
  - Gaithersburg, Maryland
  - Boston, Massachusetts
  - Gardner, Massachusetts
  - North Dartmouth, Massachusetts
  - Taunton, Massachusetts
  - Liberty, Missouri
  - Sasint Louis, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Bellevue, Nebraska
  - Omaha, Nebraska
  - Cranford, New Jersey
  - Edison, New Jersey
  - Hillsborough, New Jersey
  - Verona, New Jersey
  - Albany, New York
  - Middletown, New York
  - Mineola, New York
  - Mount Vernon, New York
  - New Paltz, New York
  - New York, New York
  - Newburgh, New York
  - Olean, New York
  - Rockville Centre, New York
  - Staten Island, New York
  - The Bronx, New York
  - Asheville, North Carolina
  - High Point, North Carolina
  - Fargo, North Dakota
  - Beavercreek, Ohio
  - Centerville, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Altoona, Pennsylvania
  - Beaver, Pennsylvania
  - Carlisle, Pennsylvania
  - Harrisburg, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Upland, Pennsylvania
  - Lincoln, Rhode Island
  - Greenville, South Carolina
  - Knoxville, Tennessee
  - Dallas, Texas
  - El Paso, Texas
  - Garland, Texas
  - Heath, Texas
  - Round Rock, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Spokane, Washington
  - Tacoma, Washington
  - Wheeling, West Virginia
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 88 | 88
Completed | 78 | 74
Not Completed | 10 | 14
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 8 | 7
Not completed — Patient Decision to Withdraw | 2 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 88 | 88 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.14 (11.73) | 51.86 (13.25) | 51.50 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 60 | 123
  Male | 25 | 28 | 53

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Not Experiencing a Protocol-defined Severe Exacerbation During the Study
Description: A protocol-defined severe exacerbation was a clinically significant worsening of asthma which, in the clinical judgment of the investigator, required at least 1 of the following: (1) Initiation of systemic corticosteroid treatment (tablets, suspension, or injection) or an increase in the level of systemic corticosteroid treatment from a stable maintenance dose for at least 3 days (For patients taking chronic oral corticosteroids, a protocol-defined severe exacerbation was any clinically significant worsening of asthma requiring ≥ 3 days of treatment with at least a 20 mg increase in the average daily dose of oral prednisone or a comparable dose of systemic corticosteroids) or (2) a hospitalization or emergency room visit because of asthma requiring systemic corticosteroids.
Time Frame: Baseline to the end of the study (up to 52 weeks)
Population: Intent-to-treat population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 88 | 88
Percentage of participants | 67.0 [57.2 to 76.9] | 47.7 [37.3 to 58.2]
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 19.3, 95% CI 2-sided [5.0 to 33.6]

2. Secondary Outcome: Time to the First Protocol-defined Severe Exacerbation
Description: as for outcome 1
Time Frame: Baseline to the end of the study (up to 52 weeks)
Population: Intent-to-treat population: All randomized participants.
Measure: Mean (95% Confidence Interval); unit: Weeks
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 88 | 88
Weeks | 21.7 [14.41 to 29.03] | 16.6 [11.90 to 21.26]

ADVERSE EVENTS:
Description: Safety population: All randomized participants who had at least 1 injection.
  Adverse events for participants who crossed-over from placebo to Xolair are included in the Xolair Continuation group. Participants randomized to placebo who switched before 52 weeks are included in both columns; their adverse events are only reported once.
Arm/Group | Omalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 10/121 | 8/88
Other Adverse Events (participants affected / at risk) | 100/121 | 88/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=121) | Placebo (N=88)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0
Dyskinesia oesophageal (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mueller's mixed tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Haematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=121) | Placebo (N=88)
Bronchitis (Infections and infestations) | 9 | 8
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 26 | 12
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 23 | 11
Urinary tract infection (Renal and urinary disorders) | 6 | 6
Asthma (Immune system disorders) | 28 | 30
Rhinitis allergic (Immune system disorders) | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.